CLINICAL TRIAL: NCT01478880
Title: Efficacy and Safety of Bilateral Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation) for the Treatment of Auditory Hallucinations
Brief Title: Efficacy and Safety of Bilateral Theta Burst Stimulation for the Treatment of Auditory Hallucinations
Acronym: TBS-H
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBS-H 1
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Auditory Hallucinations
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cTBS (Experimental)
  Interventions: Procedure: continuous theta burst stimulation (cTBS)
- Sham cTBS (Sham Comparator)
  Interventions: Procedure: sham cTBS

INTERVENTIONS:
Procedure: continuous theta burst stimulation (cTBS) — bilateral continuous theta burst stimulation (bursts of 3 stimuli, 50Hz every 200ms for 40s, 80% active motor threshold) to the temporoparietal cortex (EEG 10/20: halfway T3/P3 and T4/P4)
  Arms: cTBS
Procedure: sham cTBS — bilateral continuous theta burst stimulation (bursts of 3 stimuli, 50Hz every 200ms for 40s, 80% active motor threshold) to the temporoparietal cortex (EEG 10/20: halfway T3/P3 and T4/P4) with the stimulation coil tilted 45°
  Arms: Sham cTBS

SUMMARY:
First clinical studies indicate an effect of repetitive transcranial magnetic stimulation(rTMS) in the treatment of auditory hallucinations (AH). However, effect size, optimal stimulation site and parameters are unclear. With this randomized, placebo-controlled clinical trial we test the efficacy and safety of bilateral continuous theta burst stimulation (cTBS), a patterned form rTMS, against auditory hallucinations. The treatment will be applied add-on to individual antipsychotic and behavioral therapy. Patients will be treated for 6 weeks each weekday (30 sessions) with 40s of cTBS (halfway between T3/P3 and T4/P4). For weeks 1-3, half of the subjects will be randomized to a sham-stimulation (coil tilted 45°). During weeks 4-6, all subjects receive real cTBS.

ELIGIBILITY:
Inclusion Criteria:

* auditory hallucinations at least once a week
* Schizophrenia (DSM-IV)
* stable treatment setting (in- or out-patient)
* no change of antipsychotics during and at least 1 week before treatment initiation

Exclusion Criteria:

* epilepsy
* benzodiazepines > 1,5mg lorazepam / d
* pregnancy
* metal parts in the brain
* cardiac pacemaker
* deep brain stimulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Psychotic Symptom Rating Scales (PSYRATS), subscale for auditory hallucinations | 3 weeks
  Change of PSYRATS AH score compared to baseline after 3 weeks of treatment

SECONDARY OUTCOMES:
Hallucination change score (HCS) | 3 and 6 weeks
Positive and Negative Symptom Scale (PANSS) | 3 and 6 weeks
PSYRATS subscale for auditory hallucinations | 6 weeks
  Change of PSYRATS AH score compared to baseline after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, MD, Principal Investigator — Universtity of Tuebingen
Locations (1):
- University of Tübingen, Department of Psychiatry and Psychotherapy, Tübingen, Germany